CLINICAL TRIAL: NCT03277703
Title: Booster Vaccine Strategy to Improve Serologic Responses to Influenza Vaccination in Children With Rheumatic Diseases and Inflammatory Bowel Disease Who Are Receiving Immunosuppressive Therapies
Brief Title: Flu Vaccine Response in Patients on Biologic Therapies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Christy Beneri, Assistant Professor of Pediatrics, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1077651
Record Dates: First submitted 2017-08-30; First posted 2017-09-11 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Rheumatologic Disorder; Inflammatory Bowel Diseases; Immune Complex Diseases
Keywords: Influenza vaccine; Booster dose; immunocompromised; Biologic therapy; Rheumatologic disease; inflammatory bowel disease
MeSH Terms: conditions — Collagen Diseases; Inflammatory Bowel Diseases; Immune Complex Diseases; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - Booster (Experimental): Group 1 subjects will receive a second booster dose of injectable influenza vaccine 4 weeks after initial vaccination in year 1 and year 2.
  Interventions: Biological: Influenza vaccine
- Group 2 - Standard (Active Comparator): Group 2 subjects will be receive the standard single dose of influenza vaccine in year 1 but will receive a second booster dose of injectable influenza vaccine 4 weeks after initial vaccination in year 2.
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — The primary aim of this study is to assess the immunogenicity of booster dose influenza vaccine strategy in patients with rheumatologic diseases and IBD who are receiving immunosuppressive therapies.
  Secondary aims of this study include assessment of the safety and clinical efficacy, of booster dose influenza vaccine in the prevention of influenza-like illnesses (ILI) in this patient population

SUMMARY:
This proposed study will assess the immunogenicity, safety, and clinical efficacy of an influenza vaccine booster dose strategy in patients with autoimmune diseases who are receiving immunosuppressive therapies. Investigators will compare serologic responses to single versus a booster dose of influenza vaccine in patients with inflammatory bowel disease (IBD- Crohn's Disease or Ulcerative Colitis) or rheumatologic diseases who are receiving immunosuppressive therapies. Subjects will be randomized to receive either one or two doses of influenza vaccination in year #1. In year# 2, all participants will be given two doses of influenza vaccine. Serologic responses will be measured pre and 4-6 weeks post vaccination. This study will also assess the immunogenicity and safety of a booster vaccine strategy in the prevention of influenza-like illness (ILI). Investigators anticipate that booster dose strategy will improve both clinical and serologic responses in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 3-22 years
* Rheumatologic condition (JIA, Uveitis, SLE and other rheumatologic disorders) or inflammatory bowel disease (Crohn's disease or ulcerative colitis) and who are receiving immunosuppressive therapies as follows:

  * TNF inhibitors [etanercept (Enbrel), adalimumab (Humira®), infliximab (Remicade®)]
  * anti IL -1 [anakinra (Kineret®) or canakinumab (Ilaris®)]
  * IL-6 tocilizumab (Actemra®)
  * anti IL-12/23 ustekinumab (Stelara®)
  * anti CTLA-4 [abatacept (Orencia®)]
  * vedolizumab (Entyvio®)
  * azathioprine (Imuran®)
  * 6 mercaptopurine (Purinethol®)
  * Cyclosporine
  * Leflunomide
  * Mycophenolate
  * methotrexate (Otrexup® or Rasuvo®)

Exclusion Criteria:

* Prior allergic reaction to any vaccine components
* Other contraindication to influenza vaccination
* Severe egg allergy
* Pregnancy
* Prior Guillain-Barre syndrome
* Therapy with oral corticosteroids ≥2 mg/mg/day within 4 weeks of study entry
* Prior rituximab
* Prior cyclophosphamide
* Prior IVIG within 8 weeks
* Acute febrile illness at time of study evaluation
* No prior history of two doses of influenza in the past for ages 3-8 years

Ages: 3 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Influenza hemagglutination inhibition (HAI) titer | 4 weeks post vaccination
  immunological vaccine response

SECONDARY OUTCOMES:
Clinical efficacy of vaccine | through study completion, an average of 2 years
  decreased influenza rates

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, East Setauket, New York, United States

REFERENCES:
- [Background] Walters HM, Pan N, Lehman TJ, Adams A, Huang WT, Sitaras L, Cunningham-Rundles S, Walsh TJ, Toussi SS. A prospective study comparing infection risk and disease activity in children with juvenile idiopathic arthritis treated with and without tumor necrosis factor-alpha inhibitors. Clin Rheumatol. 2015 Mar;34(3):457-64. doi: 10.1007/s10067-014-2779-8. Epub 2014 Sep 18. PMID 25227771
- [Background] Toussi SS, Pan N, Walters HM, Walsh TJ. Infections in children and adolescents with juvenile idiopathic arthritis and inflammatory bowel disease treated with tumor necrosis factor-alpha inhibitors: systematic review of the literature. Clin Infect Dis. 2013 Nov;57(9):1318-30. doi: 10.1093/cid/cit489. Epub 2013 Jul 29. PMID 23899685
- [Background] Carvalho LM, de Paula FE, Silvestre RV, Roberti LR, Arruda E, Mello WA, Ferriani VP. Prospective surveillance study of acute respiratory infections, influenza-like illness and seasonal influenza vaccine in a cohort of juvenile idiopathic arthritis patients. Pediatr Rheumatol Online J. 2013 Mar 7;11:10. doi: 10.1186/1546-0096-11-10. eCollection 2013. PMID 23510667
- [Background] Aikawa NE, Campos LM, Silva CA, Carvalho JF, Saad CG, Trudes G, Duarte A, Miraglia JL, Timenetsky Mdo C, Viana VS, Franca IL, Bonfa E, Pereira RM. Glucocorticoid: major factor for reduced immunogenicity of 2009 influenza A (H1N1) vaccine in patients with juvenile autoimmune rheumatic disease. J Rheumatol. 2012 Jan;39(1):167-73. doi: 10.3899/jrheum.110721. Epub 2011 Nov 15. PMID 22089462
- [Background] Flannery B, Reynolds SB, Blanton L, Santibanez TA, O'Halloran A, Lu PJ, Chen J, Foppa IM, Gargiullo P, Bresee J, Singleton JA, Fry AM. Influenza Vaccine Effectiveness Against Pediatric Deaths: 2010-2014. Pediatrics. 2017 May;139(5):e20164244. doi: 10.1542/peds.2016-4244. Epub 2017 Apr 3. PMID 28557757
- [Background] Ogimi C, Tanaka R, Saitoh A, Oh-Ishi T. Immunogenicity of influenza vaccine in children with pediatric rheumatic diseases receiving immunosuppressive agents. Pediatr Infect Dis J. 2011 Mar;30(3):208-11. doi: 10.1097/INF.0b013e3181f7ce44. PMID 20861757
- [Background] deBruyn J, Fonseca K, Ghosh S, Panaccione R, Gasia MF, Ueno A, Kaplan GG, Seow CH, Wrobel I. Immunogenicity of Influenza Vaccine for Patients with Inflammatory Bowel Disease on Maintenance Infliximab Therapy: A Randomized Trial. Inflamm Bowel Dis. 2016 Mar;22(3):638-47. doi: 10.1097/MIB.0000000000000615. PMID 26595551
- [Background] Cordero E, Roca-Oporto C, Bulnes-Ramos A, Aydillo T, Gavalda J, Moreno A, Torre-Cisneros J, Montejo JM, Fortun J, Munoz P, Sabe N, Farinas MC, Blanes-Julia M, Lopez-Medrano F, Suarez-Benjumea A, Martinez-Atienza J, Rosso-Fernandez C, Perez-Romero P; TRANSGRIPE 1-2 Study Group. Two Doses of Inactivated Influenza Vaccine Improve Immune Response in Solid Organ Transplant Recipients: Results of TRANSGRIPE 1-2, a Randomized Controlled Clinical Trial. Clin Infect Dis. 2017 Apr 1;64(7):829-838. doi: 10.1093/cid/ciw855. PMID 28362949